CLINICAL TRIAL: NCT01753063
Title: Managing Expectations in Pediatric Weight Management: A Pilot Study in Focus on a Fitter Future III Hospitals
Brief Title: Managing Patient Expectations in Pediatric Weight Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: University of Nebraska (Other); Nationwide Children's Hospital (Other); Connecticut Children's Medical Center (Other); Mt. Washington Pediatric Hospital (Unknown); C.S. Mott Children's Hospital (Other); Children's Hospital Colorado (Other); Children's Hospital of Illinois (Unknown); Helen DeVos Children's Hospital (Other); OHSU Doernbecher Children's Hospital (Other); Norton Healthcare (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: P00006045
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Obesity
Keywords: Obesity; Children; Adolescents; Attrition
MeSH Terms: conditions — Obesity; Tooth Wear | interventions — Treatment Expectations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient Expectations (Experimental): At the family's initial visit to the pediatric weight management program/clinic each parent/guardian and adolescent (if age 12 yrs. or older) will complete the survey tool. At 3 months, families will be asked to complete a follow up survey. This will be fielded at a visit for those returning to clinic or by phone/mail for those not returning.
  Interventions: Behavioral: Patient Expectations

INTERVENTIONS:
Behavioral: Patient Expectations — Baseline Expectations survey (parent/guardian and adolescents 12 and older)
Behavioral: Patient Expectations — 3 month follow up survey (parent/guardian and adolescents 12 and older)

SUMMARY:
As part of Children's Hospital Association's Focus on a Fitter Future III Obesity Task Force, this project will target patient and family expectations across the domains of nutrition, physical activity and behavior change/family support as a means of patient engagement and retention in pediatric weight management. This will be a prospective, non-randomized, uncontrolled, single-arm trial for children between 2 and 18 years of age and a parent/guardian, who are starting a pediatric weight management program/clinic in one of the participating centers. The parent/guardian and child if 12 years of age or older receive a survey at the first visit, which asks about their expectations and goals for the visit. This information will then be used as part of clinical care to tailor treatment. After 3 months, the parent/guardian and adolescent, if applicable, will receive a follow up survey asking about their progress in these areas.

ELIGIBILITY:
Inclusion Criteria:

* Subject conversant in English or Spanish
* Parent/guardian conversant in English or Spanish
* Patient aged 2-18 years

Exclusion Criteria (For Adolescent):

• Parent-reported cognitive issues preventing completion of the form, such as in-school aide>50% of the school day; special education classes >50% of school day

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 405 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Attrition at 3 months | 3 months
  Defined for treatment clinics (i.e., no set end point) as attending an initial appointment but no further appointments in a 3 month period. For treatment programs (i.e., set end point), attrition is defined as attending <25% of visits in a 3 month period

SECONDARY OUTCOMES:
Congruence of learning needs and achieved outcomes | 3 months
  Defined as a match between the identified most important treatment expectation in each of the domains at baseline and the most helpful treatment domains at 3 months. Congruent = at least 4 out 6 possible matches.

OTHER OUTCOMES:
Matched expectations between parent and child expectations at baseline | Baseline
  match between the identified most important treatment expectation in each of the domains at baseline for the parent and adolescent (age 12+). Matched= at least 4 out 6 possible matches.
Child BMI Z-score | Baseline, 3 months
  Change in BMI z-score between baseline and 3 month follow-up
Provider Satisfaction | 3 months
  Providers will complete a brief survey at the end of the recruitment phase to solicit general feedback and to assess the tool's utility and impact on clinical flow.
Participation Rate | Baseline
  Proportion of patients who enrolled among those invited to participate.

CONTACTS AND LOCATIONS:
Overall Officials: Erinn Rhodes, MD, MPH, Study Chair — Boston Children's Hospital; Sarah Hampl, MD, Study Chair — Children's Mercy Hospitals & Clinics
Locations (12):
- United States (12):
  - Children's Hospital, Colorado, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Children's Hospital of Illinois, Peoria, Illinois
  - Kosair Children's Hospital, Louisville, Kentucky
  - Mt. Washington Pediatric Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Children's Mercy Hospitals & Clinics, Kansas City, Missouri
  - Children's Hospital and Medical Center, Omaha, Omaha, Nebraska
  - Nationwide Children's Hospital, Columbus, Ohio
  - Doernbecher Children's Hospital OHSU, Portland, Oregon

REFERENCES:
- [Background] Hampl S, Demeule M, Eneli I, Frank M, Hawkins MJ, Kirk S, Morris P, Sallinen BJ, Santos M, Ward WL, Rhodes E. Parent perspectives on attrition from tertiary care pediatric weight management programs. Clin Pediatr (Phila). 2013 Jun;52(6):513-9. doi: 10.1177/0009922813482515. Epub 2013 Mar 28. PMID 23539682
- [Background] Sallinen Gaffka BJ, Frank M, Hampl S, Santos M, Rhodes ET. Parents and pediatric weight management attrition: experiences and recommendations. Child Obes. 2013 Oct;9(5):409-17. doi: 10.1089/chi.2013.0069. Epub 2013 Sep 12. PMID 24028563
- [Derived] Rhodes ET, Boles RE, Chin K, Christison A, Testa EG, Guion K, Hawkins MJ, Petty CR, Sallinen Gaffka B, Santos M, Shaffer L, Tucker J, Hampl SE. Expectations for Treatment in Pediatric Weight Management and Relationship to Attrition. Child Obes. 2017 Apr;13(2):120-127. doi: 10.1089/chi.2016.0215. Epub 2017 Jan 16. PMID 28092464